CLINICAL TRIAL: NCT03858686
Title: The Effect of FP-025, a MMP-12 Inhibitor, on Allergen-induced Airway Responses, Airway Inflammation and Aspects of Airway Remodeling in Subjects With Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma (HDM)-Allergic Asthma
Brief Title: The Effect of FP-025, on Allergen-induced Airway Responses in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: FP02C-18-001
Record Dates: First submitted 2018-08-09; First posted 2019-03-01 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Asthma, COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — FP-025

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 400 mg FP-025 capsules (Active Comparator): Based on a double-blind randomized schedule, 16 subjects will receive FP-025 capsules in Period 1 and matching placebo FP-025 capsules in Period 2. Both study periods will follow the same schedule of procedures, with a washout period of at least 3 weeks and up to 7 weeks between study periods.
  Interventions: Drug: FP-025 capsules; Drug: Placebo FP-025 capsules
- FP-025 Placebo Capsules (Placebo Comparator): Based on a double-blind randomized schedule, 16 subjects will receive matching placebo FP-025 capsules in Period 1 and FP-025 capsules in Period 2. Both study periods will follow the same schedule of procedures, with a washout period of at least 3 weeks and up to 7 weeks between study periods.
  Interventions: Drug: FP-025 capsules; Drug: Placebo FP-025 capsules

INTERVENTIONS:
Drug: FP-025 capsules — FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
  Other Names: Adermastat
Drug: Placebo FP-025 capsules — Placebo FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
  Other Names: Placebo

SUMMARY:
This study is a Phase IIa, randomized, placebo-controlled, double-blind, 2-way crossover, 2-center (conducted in EU; The Netherlands) study in male and female subjects with stable, mild HDM-allergic asthma.

DETAILED DESCRIPTION:
This study is a Phase IIa, randomized, placebo-controlled, double-blind, 2-way crossover, 2-center (conducted in EU; The Netherlands) study in male and female subjects with stable, mild HDM-allergic asthma. The study will consist of two identical study periods of 12 treatment days each, separated by a washout period of at least 3 weeks (and no more than 7 weeks). Approximately 36 eligible subjects will be enrolled, to yield 32 evaluable subjects who will be treated with both FP-025 (400 mg BID) or matching placebo in a cross-over design from the evening of Day 1 till the morning of Day 12 (22 doses per study period in total).

ELIGIBILITY:
Inclusion Criteria:

The following criteria must be met by all subjects considered for study participation:

1. Females or males, between 18 and 55 years of age at Screening, inclusive, on the day of signing the Informed Consent Form (ICF).
2. Apart from a clinically stable asthma and HDM-allergy, subjects should be generally healthy with no history of a clinically relevant medical condition that in the opinion of the investigator might interfere with successful study conduct and no clinically relevant abnormalities on medical history, physical exam, vital signs, laboratory parameters or ECG at Screening.
3. Subject has a BMI ≥ 18.0 kg/m2 and ≤ 32.0 kg/m2 (and weighs ≥50 kg).
4. Subjects have been diagnosed with asthma cf GINA guidelines.
5. Subjects should have established allergy for HDM (serum HDM-specific IgE or positive SPT at Screening or documented within 1 year pre-screening).
6. No severe exacerbation of asthma within past 1 year requiring hospital admission and/or treatment with oral corticosteroids; no (never) intensive care admissions for asthma or intubation).
7. FEV1 should be ≥70% of predicted on Screening Day 2.
8. On Screening Day 2, PC20FEV1(Meth) should be <16 mg/mL if methacholine chloride is used (or adjusted by a factor of 1.2 if methacholine bromide is used).
9. Baseline blood eosinophils should be ≥150 cells/μL at Screening or documented within 3 months before Screening Day 1.
10. Subjects should have a documented airway late response to inhaled HDM on Screening Day 3.
11. Subjects of childbearing potential must be willing to use adequate contraception (double-barrier) or must refrain from intercourse.
12. Female subjects of non-childbearing potential must have had

    ≥ 12 months of spontaneous amenorrhea (with folliclestimulating hormone [FSH] ≥ 30 mIU/mL). Surgically sterile women are defined as those who have had a hysterectomy, bilateral ovariectomy (for 'benign' reasons), or bilateral tubal ligation.
13. All female subjects should have a negative pregnancy test at Screening and on Day -1.
14. Negative alcohol breath test on Screening Day 1 and Day -1.
15. Negative cotinine test on Screening Day 1 and Day -1.
16. Negative urine drug screen for recreational and other drugs on Screening Day 1 and Day -1.
17. Subjects are non-smokers. A non-smoker is defined as an individual who has abstained from smoking for at least 1 year prior to Screening Day 1. Number of years smoked x number of packs per day should be <5 pack years.
18. Subject should be willing and able to perform the lung function tests and other study-related procedures and comply with study protocol requirements.
19. Subject should provide a signed and dated informed consent.

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

1. Subject has any active and/or chronic (physical or mental) condition requiring maintenance (pharmaco)therapy or which otherwise precludes subject from safe or adequate study participation (ineligibility will be assessed by the PI).
2. Subject has a history of cancer (exception: localized basalioma or cervix carcinoma in situ).
3. Subject had any major (nasal) surgery in the 6 months before Screening Day 1.
4. Subject is pregnant or lactating.
5. Subject is using immunotherapy that according to the PI may interfere with the study (e.g. in case of immunotherapy with HDM or when subject is in the updosing phase of any immunotherapy).
6. Subject regularly used alcohol (intake of >21 units/wk for males and >14 units/wk for females) and/or recreational drugs within the last 6 months prior to screening.
7. Subject had any respiratory (viral) infections (e.g. common cold) within 3 weeks of Screening Day 1 or on Day -1.
8. Subject is using maintenance asthma therapy or long-acting bronchodilators or any other anti-asthma or anti-allergic medications (as detailed in the protocol) other than infrequent use of SABA prn only.
9. Subject is using prohibited medications as detailed in the protocol.
10. Multi-sensitized symptomatic subjects with seasonal (pollen) allergies should be included outside of the relevant allergen season and/or should not be in frequent contact with the relevant allergen during the study.
11. Subject has any known allergic response for the medications used or known severe allergic reactions or anaphylaxis (to food/medications/insect venoms).
12. Subject participated in medical studies in the past 3 months (non-biologicals) or in the past 6 months (biologicals).
13. Subject is anticipated not to comply with study medication or other aspects of the study (at the discretion of the investigator).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Diamant, MD, PhD, Principal Investigator — QPS Netherlands; Rene Lutter, Principal Investigator — Academic Medical Centre/University of Amsterdam
Locations (2):
- Netherlands (2):
  - Academic Medical Centre/University of Amsterdam, Department of Respiratory Medicine and Experiment Immunology, Amsterdam
  - QPS Netherlands - Clinical Pharmacology Unit, Groningen

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FP-025 - Placebo: Based on a double-blind randomized schedule, subjects will receive FP-025 capsules BID in Period 1 and matching placebo capsules BID in Period 2.
  Both study periods will follow the same schedule of procedures, with a washout period of at least 3 weeks and up to 7 weeks between study periods.
- Placebo - FP-025: Based on a double-blind randomized schedule, subjects will receive matching placebo capsules BID in Period 1 and FP-025 capsules BID in Period 2.
  Both study periods will follow the same schedule of procedures, with a washout period of at least 3 weeks and up to 7 weeks between study periods.
Period: Period 1
Arm/Group | FP-025 - Placebo | Placebo - FP-025
Started | 13 | 14
Completed | 12 | 11
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Lack of compliance | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout
Arm/Group | FP-025 - Placebo | Placebo - FP-025
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Period 2
Arm/Group | FP-025 - Placebo | Placebo - FP-025
Started | 12 | 11
Completed | 12 | 10
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FP-025 - Placebo: Based on a double-blind randomized schedule, 16 subjects will receive FP-025 capsules in Period 1 and matching placebo FP-025 capsules in Period 2. Both study periods will follow the same schedule of procedures, with a washout period of at least 3 weeks and up to 7 weeks between study periods.
  FP-025 capsules: FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
  Placebo FP-025 capsules: Placebo FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
- Placebo - FP-025: Based on a double-blind randomized schedule, 16 subjects will receive matching placebo FP-025 capsules in Period 1 and FP-025 capsules in Period 2. Both study periods will follow the same schedule of procedures, with a washout period of at least 3 weeks and up to 7 weeks between study periods.
  FP-025 capsules: FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
  Placebo FP-025 capsules: Placebo FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
- Total: Total of all reporting groups
Arm/Group | FP-025 - Placebo | Placebo - FP-025 | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (6.22) | 26.9 (7.3) | 26.9 (6.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Netherlands | 13 | 14 | 27
FEV1 % predicted [Mean (Standard Deviation); unit: % predicted] | 88.95 (8.26) | 92.04 (13.3) | 90.44 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Effect of FP-025 Versus Placebo on the Allergen (HDM)-Induced Late Asthmatic Response (LAR) in Subjects With Clinically Stable, Mild Allergic Asthma and Blood Eosinophilia.
Description: Late asthmatic response (LAR) is defined as FEV1 AUC3-8h; differences between FP025 and placebo in subjects with clinically stable, mild allergic asthma and blood eosinophilia.
Time Frame: FEV1 measured hourly from 3 to 8 hours post dose on Day 11 During Placebo and FP-025 in Subjects with HDM-Allergic Mild Asthma with Blood Eosinophilia to generate LAR(AUC3-8h)
Population: Of the total 22 subjects who completed both periods 3 were not included in the final analysis: 1 in the FP-025-placebo sequence due to poor PFT variability throughout trial periods, 2 in the placebo-FP-025 sequence due to high deviation in the PC20FEV1(Meth) test results between period 1 and period 2. In addition, carry-over effect was detected in the period 2(placebo) data for FP-025-placebo sequence. Thus the final subjects analyzed include 19 FP-025 treated and 8 placebo treated patients.
Measure: Mean (Standard Deviation); unit: h*%
Groups:
- FP-025: Based on a double-blind randomized schedule, 16 subjects will receive FP-025 capsules in Period 1 and matching placebo FP-025 capsules in Period 2. Both study periods will follow the same schedule of procedures, with a washout period of at least 3 weeks and up to 7 weeks between study periods.
  FP-025 capsules: FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
  Placebo FP-025 capsules: Placebo FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
- Placebo: Based on a double-blind randomized schedule, 16 subjects will receive matching placebo FP-025 capsules in Period 1 and FP-025 capsules in Period 2. Both study periods will follow the same schedule of procedures, with a washout period of at least 3 weeks and up to 7 weeks between study periods.
  FP-025 capsules: FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
  Placebo FP-025 capsules: Placebo FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
h*% | -80.33 (47.33) | -113.43 (48.6)

2. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in Late Asthmatic Response (LAR)
Description: Late asthmatic response (LAR) expressed as max% fall in FEV1 from post-diluent 3-8 h(LAR) baseline post allergen challenge in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Maximal percentage fall
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
Maximal percentage fall | -27.716 (14.3153) | -36.605 (15.0187)

3. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in EAR.
Description: Early asthmatic response (EAR) expressed as FEV1 AUC0-3h in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma.
Time Frame: FEV1 measured hourly from 0 to 3 hours post dose on Day 11 During Placebo and FP-025 in Subjects with HDM-Allergic Mild Asthma with Blood Eosinophilia to generate EAR(AUC0-3h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*%
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
h*% | -35.748 (26.2807) | -28.683 (25.4041)

4. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in Early Asthmatic Response (EAR).
Description: Early asthmatic response (EAR) expressed as max% fall in FEV1 from post-diluent 0-3 h(EAR) baseline post allergen in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma.
Time Frame: FEV1 measured hourly from 0 to 3 hours post dose on Day 11 During Placebo and FP-025 in Subjects with HDM-Allergic Mild Asthma with Blood Eosinophilia to generate maximal% fall in FEV1(0-3h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Maximal percentage fall
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
Maximal percentage fall | -26.070 (14.2299) | -20.294 (14.5720)

5. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in Joint HDM-induced Airway Response.
Description: Joint HDM-induced airway response expressed as FEV1 AUC0-8h post-allergen in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma patients.
Time Frame: FEV1 measured hourly from 0 to 8 hours post dose on Day 11 During Placebo and FP-025 in Subjects with HDM-Allergic Mild Asthma with Blood Eosinophilia to generate FEV1(AUC0-8h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*%
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
h*% | -117.543 (67.4201) | -141.166 (54.9937)

6. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in Airway Hyper-responsiveness
Description: Changes in allergen-induced AHR: i.e: PC20FEV1(Meth) or PC20FEV1(Hist) pre-post allergen (Day 10 versus Day12) in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma.
Time Frame: PC20FEV1(Meth) or PC20FEV1(Hist) measured pre and post allergen (Day 10 versus Day12 in period 1 and period 2) in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
mg/mL | 0.460 (3.4385) | 0.282 (3.1754)

7. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in Small Airway Parameters Following HDM-challenge, IOS R5 (AUC3-8 Hours)
Description: Small airway parameters measured by IOS R5(AUC3-8h) during LAR post-allergen challenge in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Time Frame: IOS R5 measured hourly from 3 to 8 hours post dose on Day 11 During Placebo and FP-025 in Subjects with HDM-Allergic Mild Asthma with Blood Eosinophilia to generate IOS R5(AUC3-8h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*%
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
h*% | 186.438 (113.2697) | 295.400 (178.9532)

8. Secondary Outcome: The Effect of Study Treatments on Allergen (HDM)-Induced Changes in Blood Eosinophils, Day 10 vs Day 12.
Description: Changes in allergen-induced airway and systemic biomarkers (i.e. eosinophils (blood) (Day 10 versus Day12) (potential treatment effect).
Time Frame: Blood eosinophils measured pre and post allergen (Day 10 versus Day12 in period 1 and period 2) in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 Eosinophils/L
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
10^9 Eosinophils/L | 0.1061 (0.12225) | 0.1846 (0.12272)

9. Secondary Outcome: To Determine the Treatment Effect (FP-025 Versus Placebo) on Baseline Parameters (i.e. Day 1 Versus Day 10), Through Measurement of PC20FEV1.
Description: Changes in PC20FEV1(Meth) or PC20FEV1(Hist) Day 1 versus Day 10 (potential treatment effect) in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma.
Time Frame: PC20FEV1(Meth) or PC20FEV1(Hist) measured pre-allergen (Day 1 versus Day10 in period 1 and period 2) in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
mg/mL | 0.855 (2.3187) | 1.030 (2.0795)

10. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in Small Airway Parameters Following HDM-challenge, IOS R20.
Description: Small airway parameters measured by IOS R20(AUC3-8h)) during LAR post-allergen challenge in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Time Frame: IOS R20 measured hourly from 3 to 8 hours post dose on Day 11 During Placebo and FP-025 in Subjects with HDM-Allergic Mild Asthma with Blood Eosinophilia to generate IOS R20(AUC3-8h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*%
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
h*% | 62.356 (51.4601) | 98.653 (88.7628)

11. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in Small Airway Parameters Following HDM-challenge, IOS R5 - R20.
Description: Small airway parameters measured by IOS R5-R20(AUC3-8h)) during LAR post-allergen challenge in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Time Frame: IOS R5-R20 measured hourly from 3 to 8 hours post dose on Day 11 During Placebo and FP-025 in Subjects with HDM-Allergic Mild Asthma with Blood Eosinophilia to generate IOS R5-R20(AUC3-8h)
Population: Of the total 22 subjects who completed both periods 3 were not included in the final analysis: 1 in the FP-025-placebo sequence due to poor PFT variability throughout trial periods, 2 in the placebo-FP-025 sequence due to high deviation in the PC20FEV1(Meth) test results between period 1 and period 2. In addition, carry-over effect was detected in the period 2(placebo) data for FP-025-placebo sequence. Thus the final subjects analyzed include 17 FP-025 treated and 6 placebo treated patients.
Measure: Mean (Standard Deviation); unit: h*%
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 17 | 6
h*% | 1316.841 (2135.0733) | 1120.347 (339.5966)

12. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in Small Airway Parameters Following HDM-challenge, IOS AX.
Description: Small airway parameters measured by IOS Ax(AUC3-8h) during LAR post-allergen challenge in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Time Frame: IOS Ax measured hourly from 3 to 8 hours post dose on Day 11 During Placebo and FP-025 in Subjects with HDM-Allergic Mild Asthma with Blood Eosinophilia to generate IOS R5-R20(AUC3-8h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*%
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
h*% | 1641.804 (1338.5357) | 4446.304 (6444.0241)

13. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in Small Airway Parameters Following HDM-challenge, IOS X5.
Description: Small airway parameters measured by IOS X5(AUC3-8h) during LAR post-allergen challenge in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Time Frame: IOS X5 measured hourly from 3 to 8 hours post dose on Day 11 During Placebo and FP-025 in Subjects with HDM-Allergic Mild Asthma with Blood Eosinophilia to generate IOS X5(AUC3-8h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*%
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
h*% | 403.640 (237.8958) | 697.189 (807.5676)

14. Secondary Outcome: Pharmacodynamic Endpoints Include the Effect of Study Treatments on Allergen (HDM)-Induced Changes in Small Airway Parameters Following HDM-challenge, IOS FRES.
Description: Small airway parameters measured by IOS Fres(AUC3-8h) during LAR post-allergen challenge in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Time Frame: IOS Fres measured hourly from 3 to 8 hours post dose on Day 11 During Placebo and FP-025 in Subjects with HDM-Allergic Mild Asthma with Blood Eosinophilia to generate IOS Fres(AUC3-8h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*%
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
h*% | 243.149 (204.2451) | 407.199 (314.7058)

15. Other Pre Specified Outcome: To Determine the Treatment Effect (FP-025 Versus Placebo) on Baseline Parameters (i.e. Day 1 Versus Day 10) , Through Measurement of Fractionated Nitric Oxide (FeNO).
Description: FeNO is measured from exhaled air by Niox Vero® device (Circassia, Oxford, United Kingdom) according to guidelines in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma.
Time Frame: FeNO measured pre allergen (Day 1 versus Day10 in period 1 and period 2) in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
ppb | -8.12 (19.258) | -1.96 (7.712)

16. Other Pre Specified Outcome: To Determine the Treatment Effect (FP-025 Versus Placebo) on Baseline Parameters (i.e. Day 10 Versus Day 12), Through Measurement of Fractionated Nitric Oxide (FeNO).
Description: as for outcome 15
Time Frame: FeNO measured pre and post allergen (Day 10 versus Day12 in period 1 and period 2) in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
ppb | 44.94 (29.952) | 67.13 (41.906)

17. Secondary Outcome: The Effect of Study Treatments on Allergen (HDM)-Induced Changes in Blood Eosinophils, Day 1 vs Day 10.
Description: Changes in allergen-induced airway and systemic biomarkers (i.e. eosinophils (blood) (Day 1 versus Day 10) (potential treatment effect).
Time Frame: Blood eosinophils measured pre allergen (Day 1 versus Day10 in period 1 and period 2) in Mild Eosinophilic House Dust Mite (HDM)-Allergic Asthma
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 Eosinophils/L
Arm/Group | FP-025 | Placebo
Number analyzed (Participants) | 19 | 8
10^9 Eosinophils/L | 0.0461 (0.09546) | 0.0211 (0.09952)

ADVERSE EVENTS:
Time Frame: Fifteen Weeks
Groups:
- FP-025: Based on a double-blind randomized schedule, subjects will receive FP-025 capsules in Period 1 and matching placebo FP-025 capsules in Period 2. Both study periods will follow the same schedule of procedures, with a washout period of at least 3 weeks and up to 7 weeks between study periods.
  FP-025 capsules: FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
  Placebo FP-025 capsules: Placebo FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
- Placebo: Based on a double-blind randomized schedule, subjects will receive matching placebo FP-025 capsules in Period 1 and FP-025 capsules in Period 2. Both study periods will follow the same schedule of procedures, with a washout period of at least 3 weeks and up to 7 weeks between study periods.
  FP-025 capsules: FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
  Placebo FP-025 capsules: Placebo FP-025 capsules, BID will be administered to subjects in either Period 1 or Period 2, and given for 12 consecutive dosing days.
Arm/Group | FP-025 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 16/23 | 12/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FP-025 (N=23) | Placebo (N=26)
Headache (Nervous system disorders) | 5 (6) | 8 (13)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Upper Abdominal Pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dry Throat (General disorders) | 2 (2) | 0 (0)
Epistaxis (General disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-09-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT03858686/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT03858686/SAP_001.pdf
  • Informed Consent Form (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT03858686/ICF_002.pdf